CLINICAL TRIAL: NCT02853682
Title: Characterization of Endothelial Dysfunction as a Function of Hyperaemia of the Brachial Artery During Cardiac Surgery
Acronym: GLYNO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2015_843_0027
Record Dates: First submitted 2016-07-07; First posted 2016-08-03 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Capillary Leak Syndrome
Keywords: glycocalyx; capillary leak syndrome
MeSH Terms: conditions — Capillary Leak Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- presence of a vascular dysfunction: plasma
  Interventions: Biological: plasma
- absence of vascular dysfunction: plasma
  Interventions: Biological: plasma

INTERVENTIONS:
Biological: plasma — assesment of glycocalyx protein

SUMMARY:
The glycocalyx is a layer of proteins and complex sugars covering the endothelium of vessels. Its role as capillary filtration control is important. In case of alteration of the glycocalyx, experimental models and some clinical studies show an increased capillary leak responsible for interstitial edema. The analysis of glycocalyx in routine care is important to guide volume expansion. Indeed, the literature provides evidence about the poor prognosis of excess water and its impact on organ. This analysis challenge is to justify filling solution of choice according to the characteristic of this capillary leakage.

DETAILED DESCRIPTION:
Extra corporeal circulation and aortic clamp induce ischemia-reperfusion damages.

Vascular damages are represented by first glycocalyx, a layer of endovascular vessel proteoglycans, responsible for fluid permeability and secondly by nitro oxygen liberation responsible for vascular tonus.

The investigators suppose that both functions are impaired after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* cardiac surgery

Exclusion Criteria:

* auricular fibrillation
* endocarditis
* aortic dissection
* end stage chronic renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients going for cardiac surgery enrolled for 48 hours after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
glycocalyx proteins 1 | 48 hours
  proteoglycan in patient plasma is assayed.

CONTACTS AND LOCATIONS:
Overall Officials: Osama ABOU ARAB, MD, Principal Investigator — CHU Amiens; Emmanuel LORNE, MD-PhD, Study Director — CHU Amiens; Pierre-Gregoire GUINOT, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Background] Becker BF, Jacob M, Leipert S, Salmon AH, Chappell D. Degradation of the endothelial glycocalyx in clinical settings: searching for the sheddases. Br J Clin Pharmacol. 2015 Sep;80(3):389-402. doi: 10.1111/bcp.12629. Epub 2015 May 22. PMID 25778676
- [Background] Chawla LS, Ince C, Chappell D, Gan TJ, Kellum JA, Mythen M, Shaw AD; ADQI XII Fluids Workgroup. Vascular content, tone, integrity, and haemodynamics for guiding fluid therapy: a conceptual approach. Br J Anaesth. 2014 Nov;113(5):748-55. doi: 10.1093/bja/aeu298. Epub 2014 Sep 17. PMID 25231767